CLINICAL TRIAL: NCT01090219
Title: Morphofunctional Evaluations of Heavyweight and Ultralightweight Polypropylene Meshes in Men Inguinal Hernia Repair
Brief Title: Polypropylene Meshes in Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade do Extremo Sul Catarinense - Unidade Academica de Ciecias da Saude (Other)
Responsible Party: Morphofunctional evaluations of heavyweight and ultralightweight polypropylene meshes in men inguinal hernia repair, Universidade do Extremo Sul Catarinense
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0002.0.379.174.08
Record Dates: First submitted 2010-03-18; First posted 2010-03-19 (Estimated); Last update posted 2010-03-19 (Estimated); Status verified 2008-02

CONDITIONS: Inguinal Hernias
Keywords: Inguinal Hernia; contraction of two different meshes in the repair of inguinal hernias in men
MeSH Terms: conditions — Hernia, Inguinal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- two differents meshes (Experimental): Heavy-weight versus low-weight polypropylene meshes
  Interventions: Procedure: two different meshes in the repair of inguinal hernias

INTERVENTIONS:
Procedure: two different meshes in the repair of inguinal hernias — A Lichtenstein tension-free hernia repair was accomplished by emplacing Heavy-weight versus low-weight polypropylene meshes for repair of incisional hernia, marked next to the lips with six titanium clips (LT200)

SUMMARY:
The aim of this study was to analyze the shrinkage of two different screens in the repair of inguinal hernias in men . 32 patients with unilateral inguinal hernia were assigned randomly. A Lichtenstein tension-free hernia repair was accomplished by emplacing heavy weight versus ultralight weight polypropylene meshes for repair of incisional hernia, marked next to the lips with six titanium clips (LT200).

DETAILED DESCRIPTION:
eligibility criteria : Elective Surgery, men with unilateral inguinal hernia, 20 - 50 years Exclusion criteria: BMI> 30, recurrent inguinal hernia, strangulated inguinal hernia, anesthetic risk ASA III and IV, Diabetics, COPD, benign prostatic hypertrophy,cancer disease

outcome: Percentage of contraction of the different meshes by digital radiography in post-surgical days: 1, 30, 60 and 90

Independent variables: age, BMI, smoking, ethnicity, profession

ELIGIBILITY:
Inclusion Criteria:

* Elective Surgery
* Men with unilateral inguinal hernia
* Age 20 - 50 years

Exclusion Criteria:

* BMI> 30
* Recurrent inguinal hernia
* Strangulated inguinal hernia
* Anesthetic risk ASA III and IV
* Diabetics
* COPD
* Benign prostatic hypertrophy

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2008-02; Primary Completion 2010-02 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
contraction of two different meshes in the repair of inguinal hernias in men | digital radiography in post-surgical days: 1, 30, 60 and 90

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - São José Hospital, Criciúma, Santa Catarina
  - Universidade do Extremo Sul Catarinense, Criciúma, Santa Catarina